CLINICAL TRIAL: NCT06007755
Title: Exploring of Serum Biomarkers of Delirium After Cardiovascular Surgery
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Associate Professor, Huazhong University of Science and Technology
Other Study IDs: TJMZK202301
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Delirium
Keywords: delirium; biomarker; cardiovascular surgery; H3K18la; exosome; phospho-tau; Aβ
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium is determined by 3D-CAM score
- No delirium is determined by 3D-CAM score

SUMMARY:
The incidence of postoperative delirium in patients after cardiovascular surgery is very high, which seriously affects the short-term and long-term prognosis of patients, but its mechanism is not clear. Recent studies have found that lactic acid participates in the process of sepsis by inducing histone lactatation in macrophages. histone H3 lysine 18 lactylation (H3K18la) is significantly associated with the severity of disease and inflammatory response. Inflammation plays an important role in postoperative delirium. We therefore hypothesized that macrophage H3K18la also plays a role in postoperative delirium. At the same time, the latest literature shows that the early markers of Alzheimer's disease (AD), such as Aβ, exosomes and phosphorylated tau, etc. [5], can also be detected in the serum of AD patients. Given the obvious correlation between Alzheimer's disease and postoperative delirium [6], we hypothesized that serum biomarkers of AD could also be used as serum biomarkers for postoperative delirium.

The objectives of this study were to investigate the correlation between H3K18 in serum monocytes and postoperative delirium and its severity in patients undergoing cardiovascular surgery. Meanwhile, we also detect the serum levels of biomarkers of AD, such as Aβ, tau and exosomes etc., in patients undergoing major cardiac surgery. We aim to find the serum biomarkers of delirium after major cardiac surgery, so as to provide a more convenient diagnostic basis for the prevention of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

patients who receive cardiovascular surgery

* Patients participated voluntarily and signed informed consent

Exclusion Criteria:

* past medical history of neurological and psychiatric diseases; severe visual or hearing impairment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years undergoing cardiovascular surgery
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | After surgery through to postoperative day 7
  The incidence of postoperative delirium was determined according to the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) diagnostic algorithm. The algorithm consists of four clinical criteria: (1) acute onset and fluctuating course, (2) inattention, and either, (3) disorganized thinking, or(4) altered level of consciousness. To define a patient as having delirium, both the first and the second criteria have to be present, as well as either the third or the fourth criteria.

SECONDARY OUTCOMES:
the level of H3K18 in serum monocytes of postoperative delirium and un-delirium patients | Perioperative data
  Lactylation levels of all proteins and H3K18 from peripheral blood mononuclear (PBMC) were determined by western blotting and serum levels of inflammatory cytokines by flow cytometry.
the level of Aβ in serum of postoperative delirium and un-delirium patients | Perioperative data
  the level of Aβ in serum was determined by colorimetric and surface-enhanced Raman scattering (SERS) dual-mode magnetic immunosensor
the level of tau in serum of postoperative delirium and un-delirium patients | Perioperative data
  the level of tau in serum was determined by colorimetric and surface-enhanced Raman scattering (SERS) dual-mode magnetic immunosensor
the level of exosomes in serum of postoperative delirium and un-delirium patients | Perioperative data
  the level of exosomes in serum was determined by colorimetric and surface-enhanced Raman scattering (SERS) dual-mode magnetic immunosensor

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China